CLINICAL TRIAL: NCT01694654
Title: Epidemiology and Outcome of Solitary Fibrous Tumors of the Pleura. A Multicenter Study.
Brief Title: Epidemiology and Outcome of Solitary Fibrous Tumors of the Pleura.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SFT-1
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Solitary Fibrous Tumors of the Pleura

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor specimen (operative resectate)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. To determine the incidence, prevalence and long-term outcome of patients with SFTP in the German spoken part of Switzerland.
2. To define the role of immunohistochemical and molecular techniques, such as immunostaining, FISH and mutational analysis regarding their ability to predict malignant behavior in terms of prediction of overall survival and disease-free survival.

DETAILED DESCRIPTION:
Retrospective observational study on patients with SFPT in the German spoken part of Switzerland between 2000 and 2011 (approximately 300 patients):

Phase 1) Information leaflet (letter of invitation) from study center (University Hospital of Zurich) to the institutes for pathology from all university, cantonal and city hospitals in the German spoken part of Switzerland. Patient recruitment performed by medical staff from the aforementioned institutes for pathology.

Phase 2) Obtaining first orally (by telephone) and thereafter written informed consent from the patients performed by medical staff from the aforementioned institutes for pathology.

Phase 3) After written and oral consent has been given, a doctoral candidate (member of the study group, student of the University of Zurich) will perform the data entry based on clinical and histological records locally at each external institute for pathology (no patient record files will be copied or transferred in original to the University Hospital of Zurich). Data entry in the electronic case report from (excel file on study laptop) will be performed with anonymous data only. Hence, each patient will have a study number containing the treating hospital, year of diagnosis and a consecutive number (e.g. KSSG-2011-1, KSSG-2011-2, STZ-2007-1, STZ-2007-2, …). No names or birth dates will appear in the case report form.

Provided that informed consent is given, patient follow-up will be performed by contacting the primary care physician (general physician or family doctor) by telephone, which is handled by the doctoral candidate.

Deceased patients will not be incorporated within the study.

Phase 4) Review of the histological specimen which are collected by the aforementioned doctoral candidate and brought to the University Hospital of Zurich, Institute for Pathology, where immunohistochemical/molecular examinations, such as immunostaining, fluorescence in situ hybridization (FISH) and mutational analysis of the histological specimen are performed by PD Dr. A. Soltermann, member of the study team. After this, the specimens are returned to the original institute for pathology, where they were taken. All specimens are made anonymous at the moment of collection at the external hospital by the doctoral candidate (each specimen is labeled with the aforementioned study number, which is assigned in the case report form).

Phase 5) Data analysis, publication.

ELIGIBILITY:
Inclusion criteria:

* Histologically proven diagnosis of SFTP between 2000 and 2011.

Exclusion criteria:

* Missing informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Histologically proven diagnosis of SFTP between 2000 and 2011.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Divison of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Diebold M, Soltermann A, Hottinger S, Haile SR, Bubendorf L, Komminoth P, Jochum W, Grobholz R, Theegarten D, Berezowska S, Darwiche K, Oezkan F, Kohler M, Franzen DP. Prognostic value of MIB-1 proliferation index in solitary fibrous tumors of the pleura implemented in a new score - a multicenter study. Respir Res. 2017 Dec 16;18(1):210. doi: 10.1186/s12931-017-0693-8. PMID 29246159